CLINICAL TRIAL: NCT06754865
Title: A Muulticenter, Open, Non-interventional, Retrospective Cohort Study to Evaluate the Clinical Value and Safety of Xiyanping Injection in the Treatment of Acute Exacerbation of Chronic Obstructive Pulmonary Disease(COPD) Based on Real-world Clinical Data
Brief Title: Study to Evaluate the Clinical Value and Safety of Xiyanping Injection in the Treatment of Acute Exacerbation of Chronic Obstructive Pulmonary Disease(COPD) Based on Real-world Clinical Data
Acronym: XYP-202401
Status: Not yet recruiting | Type: Observational
Sponsor: Jiangxi Qingfeng Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2024XLA207-1
Record Dates: First submitted 2024-12-15; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Keywords: Acute exacerbation of chronic obstructive pulmonary disease; Xiyanping injection
MeSH Terms: interventions — Anti-Bacterial Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Exposure group: Xiyanping injection + Antimicrobial agents treatment
  Interventions: Drug: Xiyanping injection+ antibiotic
- Non-exposure group: Antimicrobial agents treatment
  Interventions: Drug: Antibiotic

INTERVENTIONS:
Drug: Xiyanping injection+ antibiotic — Xiyanping injection+ antibiotic
  Groups: Exposure group
Drug: Antibiotic — Antibiotic
  Groups: Non-exposure group

SUMMARY:
The primary objective is to evaluate the effect of Xiyanping injection on the treatment course of intravenous antibiotics for acute exacerbation of chronic obstructive pulmonary disease based on real-world clinical data, and to provide guidance and basis for the clinical application of Xiyanping injection combined with antibiotics in the treatment of acute exacerbation of chronic obstructive pulmonary disease.The secondary objectives is to evaluate the effect of Xiyanping injection on the indicators of acute exacerbation of inflammation and symptom improvement of chronic obstructive pulmonary disease.

ELIGIBILITY:
Inclusion Criteria:

1. Discharged with chronic obstructive pulmonary disease;
2. Hospitalized patients with COPD or AECOPD combined with lower respiratory tract infection;
3. The treatment course of Xiyanping injection in the exposed group was ≥3 days, and the non-exposed group did not use Xiyanping injection;
4. Study patients with complete medical records.

Exclusion Criteria:

1. Researchers believe that multiple proprietary Chinese medicines with the same or similar functions (such as Tanreqing injection, Reduning injection, Yanhuning injection, etc.) have been used at the same time during treatment, resulting in no assessment of efficacy or safety;
2. Patients with viral pneumonia or other systemic infection (such as urinary tract infection);
3. Patients who do not use intravenous antibiotics;
4. Refuse the case to be used by researchers.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with acute exacerbation of chronic obstructive pulmonary disease
Sampling Method: Non-Probability Sample
Enrollment: 1140 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Course of intravenous antibiotics | baseline, at 3(±1), 7(±1), and 10 days during medication
  Duration of intravenous antibiotic use